CLINICAL TRIAL: NCT06575621
Title: Re-imagining Hip and Knee Arthroplasty Wait-list in Nova Scotia: Pre-surgery Support Program
Brief Title: Knee-hip Surgery Wait-list Support Program
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Collaborators: Acadia University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1029156-ICF-Doyle
Record Dates: First submitted 2024-08-23; First posted 2024-08-28 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Knee Arthropathy; Hip Arthropathy
Keywords: surgery; knee; hip; exercise; risk factors
MeSH Terms: conditions — Motor Activity | interventions — Allied Health Personnel

STUDY DESIGN:
Intervention Model Description: Non-randomized intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention (Experimental): Participants receive education, medical navigation and participate in a twice weekly exercise program
  Interventions: Behavioral: Support program
- Healthy control (No Intervention): Healthy controls who are not recommended any intervention.
- Unhealthy control (No Intervention): Unhealthy controls who choose not to participate in the pre-surgery support program. Will receive recommended referrals only.

INTERVENTIONS:
Behavioral: Support program — education, medical navigation, exercise
  Arms: Intervention

SUMMARY:
This project will outline a pre-surgery support program that identifies risk factors related to poor surgical outcomes and recommends actions to improve these before surgery.

The main questions this study attempts to answer are:

1. Is a formalized knee-hip pre-surgery support program feasible, measured by recruitment rate, adherence, and completion rate?
2. Does the support program improve surgical risk factors including hemoglobin A1c (HB A1C), blood pressure, hemoglobin, estimated glomerular filtration rate (eGFR), frailty score, and physical fitness and function (measured with the 2-minute step test and 30s second sit to stand test)?

Participants will participate in education, medical navigation, and exercise.

DETAILED DESCRIPTION:
Study Design

This is a non-randomized pragmatic pilot intervention study.

Participants

Up to 100 people will participate in this pilot study. A minimum of 30 participants is required, 20 in the exercise group and 5 in each control group. This would give the investigators enough data to assess the feasibility of the exercise class as well as to develop means and standard deviations (SDs) of change that could inform a power calculation for a controlled trial.

Recruitment

Eligible participants will be identified through four Valley Regional Hospital (VRH) orthopedic surgeons' wait-lists. Staff in the surgeons' offices will contact potential participants and inform them about the study. If patients indicate they are interested and willing to be contacted by study staff, the staff member will document this and inform the research coordinator via email (NS Health email to NS Health email). The research coordinator will then contact potential participants to provide more details on the study, confirm eligibility, and, if the person is willing to participate, obtain verbal consent to enroll them in the study.

Procedures

After verbal consent to enroll in the study is obtained, the research coordinator will schedule the participant for their baseline assessment. The participant will also have the option of providing an email address to receive an electronic version of the consent form so they can review it prior to the baseline assessment. At the baseline assessment, the research coordinator will review the consent form with participants, and they will be required to sign a paper copy of the consent form at this time in order to proceed with the assessment. The research coordinator will answer any questions and address any concerns participants have regarding the study. If a participant decides they no longer want to take part in the study, the research coordinator will not proceed with the assessment. After signing the consent form, participants may withdraw at any time and will not be required to provide a reason for withdrawal.

The baseline assessment will include blood pressure, height, weight, the Oxford questionnaire, Euroqol 5 dimension questionnaire 5 level version (EQ-5D-5L), Godin-Shepherd Leisure-Time Physical Activity Questionnaire, frailty screen, and questions about demographics, health behaviours including smoking and drinking, and medical history. It will also include two fitness tests- the 2-minute step test and the 30 second sit to stand test. Bloodwork for hemoglobin A1c (Hb A1c), estimated glomerular filtration rate (eGFR), and hemoglobin (Hb) may be done at this time at the hospital lab. Although this bloodwork is normally collected at the VRH Orthopedic Assessment Clinic (OAC) initial assessment, if there is not bloodwork available within the two months prior to study enrollment, it will be requested through the OAC or by Dr. Robert Doyle.

At the end of the assessment, the research coordinator will make any recommendations to the participant based on the program algorithm. When the results of the bloodwork are available, the research coordinator will follow-up with the participants via phone call with any additional recommendations. Possible recommendations include joining the study exercise program, receiving educational videos, a consultation with a dietician, receiving smoking or alcohol cessation resources, and seeing their primary care physician or a specialist in the internal medicine department. Any necessary referrals will be made through the OAC staff (for dietician consults) or Dr. Robert Doyle (for internal medicine consults).

This process will create three study groups. Participants who do not require enhanced medical support will be 'healthy controls' due to positive health indicators. These participants will still receive educational materials and any necessary referrals, but do not have any flags that require referral for enhanced support. The primary group of interest are the 'exercise group' participants who have flags identified through the algorithm and are recommended the enhanced support that includes the exercise program. All participants who do require the exercise program will be offered a spot; however, they can decline this offer and remain in the study. This will create an additional third group of participants that are 'unhealthy controls' (i.e. those that are recommended the enhanced support but decline the exercise program). Both the healthy and unhealthy control groups are valuable to include to accurately track the break-out of participants for feasibility evaluation, as well as indicate the trajectories of status indicators for healthy and unhealthy participants while on the wait list for surgery. If the participant is recommended to exercise and chooses to take part in the study exercise program, they will undergo additional screening with the research coordinator using the Physical Activity Readiness Questionnaire (PAR-Q+) to ensure they can safely participate. Any contraindications to exercise identified during the screening process such as supplemental oxygen or resting blood pressure above 200/110 will require medical clearance prior to beginning exercise.

After the baseline assessment, variables for timepoint 0 (initial assessment at OAC) will be abstracted from patients' medical records. These variables are routinely measured at initial assessments at the OAC. Abstraction will be done by the research coordinator. To ensure the correct person's information is abstracted, the research coordinator will make sure the name, and health care number on the record match the information provided by the participant.

Participants in the exercise group will attend twice weekly hour-long sessions led by the research coordinator, who is a kinesiologist. Both virtual and in-person options will be available. In-person classes will take place at Valley Regional Hospital and Acadia University Centre for Lifestyle studies and virtual classes will be delivered via Zoom. In-person sessions will be either group personal training (3-5 participants doing their own program under the supervision of the kinesiologist) or circuit classes taught by the kinesiologist. Virtual sessions will be a circuit class taught by the kinesiologist. All necessary precautions to ensure safety will be taken including emergency contact information. For both virtual and in-person programs, each session will be comprised of aerobic, resistance, balance, and flexibility exercises. Resistance exercises will target major muscle groups including quadriceps, hamstrings, gluteals, chest, back, shoulders, biceps, and core. Sessions will begin with a warm-up and will include at least one exercise targeting each of the aforementioned muscle groups. Sessions will end with a balance exercise and stretches. The instructor will modify any exercises or offer alternatives for individuals that need them. Length of the program will vary between participants based on their surgery date. They will exercise from the time they join the program until their surgery. The last planned exercise session will be within one week of participants' surgery. It is anticipated that most participants will exercise for 8-16 weeks. A minimum duration of 6 weeks of exercise is typically needed to see significant improvements in variables due to exercise.

The principal investigator or research coordinator may remove participants from the exercise program if a change in their health makes the program unsafe for them. Examples include a heart attack, stroke, or injury that substantially impacts a participant's ability to exercise safely. If this happens, the research team will discuss with the participant whether or not they wish to remain in the study and what their options are for receiving care outside the study.

All participants will undergo a second assessment approximately two weeks before surgery. This assessment will occur at the same time as their anesthetic pre-op appointment in the pre-anesthesia clinic and will include blood tests, the Oxford questionnaire, the EQ-5D-5L, Godin physical activity questionnaire, 30 second sit to stand test, 2-minute step test, and a satisfaction survey. Staff in the pre-anesthesia clinic will complete a data collection form and administer the questionnaires and fitness tests. The medical variables included in this form, including bloodwork, are routinely measured at anesthetic pre-op appointments. To assess post-op health-related quality of life and physical function, participants will complete the questionnaires and the 30 second sit to stand test again at their six-week post-op appointment with their surgeon. Staff in the surgeon's office will complete a data collection form.

Data Analysis

Data will be cleaned prior to analysis and all variables will be examined for missing responses. Descriptive analyses will be performed for all variables to examine the distribution and outliers for the sample. All continuous variables will be examined for normal distributions by comparing the mean, SD, median, interquartile range (IQR), skewness and examining histograms. For categorical variables, frequencies and percentages will be examined.

To evaluate feasibility, recruitment rate, mean attendance to the exercise program, and completion rate will be calculated and reported. Post-op morbidity and death or serious morbidity rates and results from the satisfaction survey will also be reported. For all other outcomes, means, SDs, and 95% confidence intervals (for normally distributed data) and medians and IQR (for non-normally distributed data) will be reported. Effect sizes will be reported to inform the sample size for a future definitive trial. Program satisfaction will be assessed at follow-up using the satisfaction survey as well as semi-structured interviews with open-ended questions to understand the positive and negative aspects of each program from participants. The semi-structured interviews will be optional. These data will be analyzed in collaboration with a social scientist.

To evaluate change in risk factors, the investigators will report mean change in the questionnaires, functional, and medical/surgical outcomes. Mean change will be compared to minimally clinically important differences (MCIDs) for all outcomes which have an established MCID in hip and knee osteoarthritis patients. For outcomes which do not have an established MCID, the investigators will report the number and percentage of participants in the green, yellow and red categories at the OAC initial assessment, study baseline, and pre-surgery as well as the number and percentage of participants who move from one category to another across these three timepoints.

ELIGIBILITY:
Inclusion Criteria:

* On surgery wait list for total hip or knee arthroplasty at Valley Regional Hospital
* 18+ and able to provide informed consent
* Anticipated surgery time 8-16 weeks after the study start date

Exclusion Criteria:

* Any contraindications or exclusions identified through the assessment process that are outside thresholds for acceptable surgery risk

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-04-15 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | Study baseline
  the number of consenting participants divided by the total number of participants asked to join the study
Recruitment rate for enhanced support | Study baseline
  the number of consented and screened participants signing up to the support program, divided by the total number of participants recommended to the support program
Adherence to enhanced support program | Pre-surgery (10-16 weeks after baseline)
  percent of planned sessions attended
Completion rate | Pre-surgery (10-16 weeks after baseline)
  number of participants that completed the study divided by the number of participants that started the study

SECONDARY OUTCOMES:
Condition specific health-related quality of life | Initial assessment (approx. 6-12 months before study enrolment), study baseline, pre-surgery (10-16 weeks after baseline), post-surgery (approx. 6 weeks after surgery)
  Oxford hip/knee questionnaire, score range 12-60, lower scores are better
Generic health-related quality of life | Initial assessment (approx. 6-12 months before study enrolment), study baseline, pre-surgery (10-16 weeks after baseline), post-surgery (approx. 6 weeks after surgery)
  Euroqol 5 dimension questionnaire 5 level version (EQ-5D-5L), used to calculate health utility scores which range from 0-1, higher scores are better
Health behaviours | Study baseline and pre-surgery (10-16 weeks after baseline)
  Health behaviours questionnaire (includes questions about drinking status, number of drinks consumed per week, smoking status, and number of cigarettes smoked per day
Physical activity level | Study baseline and pre-surgery (10-16 weeks after baseline)
  Godin-Shepherd Leisure-Time Physical Activity Questionnaire (measures self-reported minutes of moderate to vigorous physical activity per week)
Physical function | Initial assessment (approx. 6-12 months before study enrolment), study baseline, pre-surgery (10-16 weeks after baseline), post-surgery (approx. 6 weeks after surgery)
  30s sit to stand test (number of repetitions completed)
Physical fitness | Study baseline and pre-surgery (10-16 weeks after baseline)
  two-minute step test (number of steps completed)
Hemoglobin A1c | Initial assessment (approx. 6-12 months before study enrolment), study baseline, pre-surgery (10-16 weeks after baseline)
  blood test
estimated glomerular filtration rate | Initial assessment (approx. 6-12 months before study enrolment), study baseline, pre-surgery (10-16 weeks after baseline)
  blood test
Hemoglobin | Initial assessment (approx. 6-12 months before study enrolment), study baseline, pre-surgery (10-16 weeks after baseline)
  blood test
Frailty | Initial assessment (approx. 6-12 months before study enrolment), study baseline, pre-surgery (10-16 weeks after baseline)
  Frailty screen, score range 1-8, lower scores are better
Body mass index | Initial assessment (approx. 6-12 months before study enrolment), study baseline, pre-surgery (10-16 weeks after baseline)
  weight and height will be combined to report BMI in kg/m^2, weight and height will be measured by research staff
Program satisfaction | Pre-surgery (10-16 weeks after baseline)
  program specific satisfaction survey
Blood pressure (systolic and diastolic) | Initial assessment (approx. 6-12 months before study enrolment), study baseline, pre-surgery (10-16 weeks after baseline)
  measured by research staff

CONTACTS AND LOCATIONS:
Overall Officials: Jonathon Fowles, PhD, Principal Investigator — Acadia University

IPD SHARING:
Plan to Share IPD: No